CLINICAL TRIAL: NCT04898920
Title: The Effect of Pre-emptive Dexamethasone on the Postoperative Analgesia After Total Hip Arthroplasty: Randomized Controlled Study
Brief Title: Pre-emptive Dexamethasone in Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 34585/3/21
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Pain
Keywords: Dexamethasone; Hip arthroplasty; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: * An anesthesia resident who will be blinded to the study groups and not participating in it will help in the preparation of uniform 10-ml syringes that contain normal saline in the control group and 16 mg dexamethasone in the other group to make the patient and care provider blinded to the group of the patient.
  * An assistant nurse who will be blinded to the study groups and will have no subsequent rule in it will help in the collection of the data of measurements to make the outcomes assessor blinded to the group of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): The patients will receive 10 ml of normal saline as a placebo dexamethasone before surgery.
  Interventions: Drug: Normal saline
- Dexamethasone Group (Experimental): Those patients will receive 16 mg dexamethasone in 10 ml of normal saline before surgery.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Normal saline — The patients will receive 10 ml of normal saline as a placebo dexamethasone before surgery.
  Other Names: Placebo
  Arms: Control Group
Drug: Dexamethasone — Those patients will receive 16 mg dexamethasone in 10 ml of normal saline before surgery.
  Other Names: Active group
  Arms: Dexamethasone Group

SUMMARY:
* Certain studies suggested that preoperative administration of systemic glucocorticoids in patients undergoing hip or knee arthroplasty surgery may improve the postoperative analgesia owing to their anti-inflammatory effect.
* This study will be carried out on 70 adult patients aged 21 to 75 years admitted to orthopedic operating rooms in Tanta university hospitals for hip surgery under spinal anesthesia. Informed written consent will be obtained from each participant.
* Patients will be randomly distributed into two equal groups using the computer-generated software.

  * Control Group: (35 patients) Those patients will receive 10 ml of normal saline before surgery.
  * Dexamethasone Group: (35 patients) Those patients will receive 16 mg dexamethasone in 10 ml of normal saline before surgery.
* Primary outcome will be postoperative morphine consumption and the secondary outcome will be the postoperative pain score

DETAILED DESCRIPTION:
- This randomized controlled prospective study will be carried out on 70 adult patients aged 21 to 75 years admitted to orthopedic operating rooms in Tanta University Hospital for hip surgery under spinal anesthesia. I

Patients will be randomly distributed into two equal groups using the computer-generated software. An anesthesia resident who will be blinded to the study groups and not participating in it will help in the preparation of uniform 10-ml syringes that contain normal saline in the control group and 16 mg dexamethasone in the other group.

* Control Group: (35 patients) Those patients will receive 10 ml of normal saline before surgery.
* Dexamethasone Group: (35 patients) Those patients will receive 16 mg dexamethasone in 10 ml of normal saline before surgery.

All the patients will undergo standardized preoperative assessment consisted of history taking, general and regional examination, and requesting preoperative investigations including (complete blood count (CBC), coagulation profile, and renal function tests). Upon patient admission to the operating theater, they will be attached to a monitor consisting of pulse oximetry, 5 lead ECG, non-invasive blood pressure, end-tidal carbon dioxide (Co2), and temperature. Then, intravenous access will be established through the insertion of an 18-gauge peripheral venous cannula, then, lactated ringer solution 7ml/kg over 30 minutes will be started. All the equipment required for spinal anesthesia, general anesthesia, and nerve block will be prepared by an expert anesthesiologist who will not be participating in this research. Also, the resuscitation equipment will be prepared before starting anesthesia.

Under complete aseptic precautions and local anesthetic skin infiltration with 3 ml lidocaine 1% at L3-L4 or L4-L5 intervertebral space, midline approach spinal anesthesia will be performed using a 25 G spinal needle. Once intrathecal placement will be confirmed, a mixture of 2 ml of hyperbaric bupivacaine (10 mg) and 0.5 ml of fentanyl (25 ugs) will be injected. The patient will be monitored for the hemodynamic parameters including the heart rate and the mean arterial pressure every 3 minutes. Moreover, the sensory and motor blockade will be assessed.

Oxygen will be applied to the patient with the aid of an oxygen mask at a flow rate of 4 L/min. The pinprick test from caudal to cephalic direction using a 26-gauge needle will be used to evaluate the sensory block until the sensory level reached the level of T11 or higher. The motor block will be assessed every 5 minutes by the Bromage score (grade 3: no movement, grade 2: unable to flex knees and can flex ankle, grade 1: unable to raise an extended leg but able to move the knees and ankles, grade 0: no paralysis) until reaching a score of 2 or 3. If no adequate sensory or motor blockade will be obtained within 20 minutes, the patient will receive general anesthesia and be excluded from the study. A decrease in the heart rate below 50 b/min will be managed by atropine 0.3 mg i.v, while a decrease in the mean arterial pressure below 65 mmHg will be managed by 10 mg ephedrine i.v and intravenous fluids.

Primary outcome will be postoperative morphine consumption and the secondary outcome will be the postoperative pain score

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA II and III, aged 21 to 75 years, admitted for hip arthroplasty surgery

Exclusion Criteria:

* Patients who refused to participate in the research
* Suspected or diagnosed coagulopathy
* Allergy to bupivacaine
* With major cardiac, renal, or hepatic disorders

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-05-23 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption | The first postoperative day
  The total dose of morphine in mg consumed in the first 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative pain score | The first postoperative day
  Postoperative Numerical Rating score (NRS) will be assessed every 2 hours in the first six hours, then every 6 hours till 24 hour.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Abdelkhalik, M.D, Principal Investigator — Tanta University
Locations (1):
- Faculty of Medicine, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data of primary outcome will be available with the corresponding author till 6 months after approval of the publication of the trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data of primary outcome will be available with the corresponding author till 6 months after approval of the publication of the trial.
Access Criteria: Contact the principal investigator